CLINICAL TRIAL: NCT03869515
Title: Genetic Causes and Clinical Features of Childhood Interstitial Lung Diseases in China
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU-02
Record Dates: First submitted 2019-02-20; First posted 2019-03-11 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Interstitial Lung Diseases of Childhood; Genetic Testing
Keywords: chILD; clinic features; genetic backgrounds; outcomes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chILD: The chILD syndrome exists when a child with DLD has had the common causes of DLD excluded as the primary diagnosis and has at least three of the following four criteria: (1) respiratory symptoms (e.g., cough, rapid and/or difficult breathing, or exercise intolerance); (2) respiratory signs (e.g., resting tachypnea, adventitious sounds, retractions, digital clubbing, failure to thrive, or respiratory fail- ure); (3) hypoxemia; and (4) diffuse abnormalities on CXR or a CT scan.
  Interventions: Other: No intervention
- Control: Healthy subjects were recruited from participants of an ongoing prospective birth cohort study: 'The Pulmonary Function Assessment for Bronchopulmonary Dysplasia (BPD) and Recurrent Lower Respiratory Tract Infections (LRTI) in Chinese Children'. Exclusion criteria were major birth defects, upper airway pathology, cardiac or neurological diseases, failure to thrive, a history of severe respiratory disease with intensive care unit admission, previous physician-diagnosed LRTI, gestational age (GA) <37 weeks or birthweight (BW) <2.5 kg.

INTERVENTIONS:
Other: No intervention — It's an observational study, so no intervention will be carried out.
  Groups: chILD

SUMMARY:
Recruitment of a carefully characterized cohort of chILD patients, to generate a database and biobank via collecting data on chILD in China. Importantly, compatibility with ongoing United States and Europe chILD data base developments will be factored in.

DETAILED DESCRIPTION:
Children Interstitial lung disease (chILD) is a heterogeneous group of rare respiratory disorders of known and unknown etiologies that are mostly chronic and associated with high morbidity and mortality. ILD are characterized by inflammatory and fibrotic changes of the lung parenchyma structure that typically result in the presence of diffuse infiltrates on lung imaging, and abnormal pulmonary function tests with evidence of a restrictive ventilatory defect and/or impaired gas exchange.

Genetic factors are important contributors to chILD. Genetic variations have been mainly described in genes encoding (or interacting with) the surfactant proteins (SP): SP-C (SFTPC) and the ATP-binding cassette-family A-member 3 (ABCA3) (ABCA3), and less frequently in the genes encoding NKX homeobox 2 (NKX2)-1 (NKX2-1), SP-B (SFTPB), SP-A (SFTPA) ,MARS and other genes.

To investigate genetic defects and clinical features of chILD in China, wide recruitment and interdisciplinary critical peer review of all diagnoses from discharge diagnosis coding system of Children's Hospital of Fudan University will be included. Each case will be given a diagnosis independently; if no firm diagnosis is possible, the investigators will review the case periodically as new information becomes available. During the first year of the study, clinicians´ decisions according to clinical practice and outcomes will be independently monitored and assessed.

The investigators will systematically optimize and clarify the relative weight of a large spectrum of single and composite clinical outcomes, sequential limited chest CT (to minimise radiation exposure), lung function testing, histopathological categorization of lung biopsies, serum markers and genetic tests. Variability, reproducibility and the effects of training on reading images will be investigated.

This project will analyse in detail treatment and outcomes within and between subjects using data collected. Analysis of the collected data will support the definition of trial protocols planned in the future.

ELIGIBILITY:
Inclusion Criteria:

* The chILD syndrome exists when a child with DLD has had the common causes of DLD excluded as the primary diagnosis and has at least three of the following four criteria: (1) respiratory symptoms (e.g., cough, rapid and/or difficult breathing, or exercise intolerance);(2) respiratory signs (e.g., resting tachypnea, adventitious sounds, retractions, digital clubbing, failure to thrive, or respiratory fail- ure); (3) hypoxemia; and (4) diffuse abnormalities on CXR or a CT scan.

Exclusion Criteria:

* These include cystic fibrosis, congenital or acquired immunodeficiency, congenital heart disease, bronchopulmonary dysplasia, pulmonary infection, primary ciliary dyskinesia presenting with newborn respiratory distress and recurrent aspiration.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: all children under 18 years old, hospitalized in Children's Hospital of Fudan University during Mar.1, 2019 and Dec.30, 2025, diagnosed with chILD , accepting empirical treatments
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosed with specific cause for chILD | 6 years
  (yes/no) Specific causes for chILD based on the 2013 Official American Thoracic Society Clinical Practice Guideline: classification, evaluation, and management of childhood interstitial lung disease in infancy

SECONDARY OUTCOMES:
Having pathogenic gene mutations | 6 years
  (yes/no) Genetic variations have been mainly described in genes encoding (or interacting with) the surfactant proteins (SP): SP-C (SFTPC) and the ATP-binding cassette-family A-member 3 (ABCA3) (ABCA3), and less frequently in the genes encoding NKX homeobox 2 (NKX2)-1 (NKX2-1), SP-B (SFTPB), SP-A (SFTPA) ,MARS and other genes.
Hypoxemia | 6 years
  (yes/no) Change of PO2 in arterial blood gases from baseline when diagnosed with chILD
Deterioration of pulmonary imaging | 6 years
  (yes/no) Change of clinical judgment on pulmonary imaging from baseline if X-ray or CT were done
Change from baseline in lung function on the spirometry forced expiratory | 6 years
  Volume at one second (FEV1) in Liter
Abnormal autoantibody at baseline when diagnosed with chILD | 6 years
  (yes/ no)
Pathological change of lung biopsy | 6 years
  (yes/no) Clinical judgment on histopathological categorization of lung biopsy when diagnosed with chILD
Deterioration of pulmonary arterial hypertension | 6 years
  (yes/no) Change of pulmonary artery pressure from baseline in echocardiagraphy
Change of BALF(bronchoalveolar lavage fluid) | 6 years
  (yes/no) Cytology analysis on BALF at the baseline when diagnosed with chILD
Survival | 1 years
  (yes/no)
Survival | 2 years
  (yes/no)
Survival | 5 years
  Five-year
Abnormal thyroid hormone at baseline when diagnosed with chILD | 6 years
  (yes/no)
Abnormal myocardial zymogram at baseline when diagnosed with chILD | 6 years
  (yes/no)
Abnormal serum immunoglobulin at baseline when diagnosed with chILD | 6 years
  (yes/no)
Abnormal serum creatinine at baseline when diagnosed with chILD | 6 years
  (yes/no)
Abnormal blood urea nitrogen at baseline when diagnosed with chILD | 6 years
  (yes/no)
Abnormal alanine transferase at baseline when diagnosed with chILD | 6 years
  (yes/no)
Abnormal allergen at baseline when diagnosed with chILD | 6 years
  (yes/no)
Recurrent hospitalization | 1 year after diagnosis
  yes:Hospitalization more than twice per year after diagnosed with chILD; no:Hospitalization less than three times per year after diagnosed with chILD;

CONTACTS AND LOCATIONS:
Overall Officials: Liling Qian, MD, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Genetic Causes, Clinical Features, Management of Childhood Interstitial Lung Diseases in China
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2019-2025
Access Criteria: Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code

REFERENCES:
- [Background] Hime NJ, Zurynski Y, Fitzgerald D, Selvadurai H, Phu A, Deverell M, Elliott EJ, Jaffe A. Childhood interstitial lung disease: A systematic review. Pediatr Pulmonol. 2015 Dec;50(12):1383-92. doi: 10.1002/ppul.23183. Epub 2015 Apr 30. PMID 25931270
- [Background] Bromley S, Vizcaya D. Pulmonary hypertension in childhood interstitial lung disease: A systematic review of the literature. Pediatr Pulmonol. 2017 May;52(5):689-698. doi: 10.1002/ppul.23632. Epub 2016 Oct 23. PMID 27774750
- [Background] Eldridge WB, Zhang Q, Faro A, Sweet SC, Eghtesady P, Hamvas A, Cole FS, Wambach JA. Outcomes of Lung Transplantation for Infants and Children with Genetic Disorders of Surfactant Metabolism. J Pediatr. 2017 May;184:157-164.e2. doi: 10.1016/j.jpeds.2017.01.017. Epub 2017 Feb 16. PMID 28215425
- [Background] Thacker PG, Vargas SO, Fishman MP, Casey AM, Lee EY. Current Update on Interstitial Lung Disease of Infancy: New Classification System, Diagnostic Evaluation, Imaging Algorithms, Imaging Findings, and Prognosis. Radiol Clin North Am. 2016 Nov;54(6):1065-1076. doi: 10.1016/j.rcl.2016.05.012. Epub 2016 Aug 12. PMID 27719976
- [Result] Kurland G, Deterding RR, Hagood JS, Young LR, Brody AS, Castile RG, Dell S, Fan LL, Hamvas A, Hilman BC, Langston C, Nogee LM, Redding GJ; American Thoracic Society Committee on Childhood Interstitial Lung Disease (chILD) and the chILD Research Network. An official American Thoracic Society clinical practice guideline: classification, evaluation, and management of childhood interstitial lung disease in infancy. Am J Respir Crit Care Med. 2013 Aug 1;188(3):376-94. doi: 10.1164/rccm.201305-0923ST. PMID 23905526